CLINICAL TRIAL: NCT04000724
Title: TechStep: Technology-based Stepped Care to Stem Transgender Adolescent Risk Transmission
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Friends Research Institute, Inc. (Other)
Collaborators: San Diego State University (Other); University of North Carolina (Other); Emory University (Other); Baylor College of Medicine (Other); Children's Hospital of Philadelphia (Other); The Fenway Institute (Other); Hunter College of City University of New York (Other); Children's Hospital Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ATN160
Record Dates: First submitted 2019-03-16; First posted 2019-06-27 (Actual); Results first posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: HIV
Keywords: Text Messaging; mHealth; HIV; AIDS; PrEP
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Text+Step (Experimental): The TechStep Text+Step messaging intervention is a six-month technology-based culturally competent theory-based text messaging intervention that sends three automated text messages to participants daily to reduce HIV risk and increase PrEP uptake and adherence.
  Interventions: Behavioral: Text Messaging (Text+Step)
- WebApp+Step (Experimental): The TechStep WebApp+Step website intervention is a six-month technology-based intervention that uses peer-to-peer interaction, daily self-monitoring, and tailored content to address barriers to HIV sexual risk reduction and PrEP uptake and adherence.
  Interventions: Behavioral: WebApp (App+Step)
- Information (Experimental): The Information/No Step intervention includes nothing more than access to a website with information about trans health, HIV/STI information and local resources tailored for transgender persons.
  Interventions: Behavioral: Information/No Step

INTERVENTIONS:
Behavioral: Text Messaging (Text+Step) — Participants receive three culturally competent, theory-based pre-written messages per day sent on a predetermined schedule. Participants who still exhibit sexual risk and do not uptake and/or adhere to PrEP at the 3-month assessment may also receive eCoaching for up to 12 weeks.
  Arms: Text+Step
Behavioral: WebApp (App+Step) — Participants receive access to a culturally competent password-protected web-based application with transgender-specific resources, support, and health information. Participants who still exhibit sexual risk and do not uptake and/or adhere to PrEP at the 3-month assessment may also receive eCoaching for up to 12 weeks.
  Arms: WebApp+Step
Behavioral: Information/No Step — Participants in the Information/No Step intervention will receive access to a static website with information about trans health, HIV/STI information and local resources tailored for transgender persons.
  Arms: Information

SUMMARY:
TechStep is a three-arm, technology-based randomized controlled trial (RCT), with a stepped care approach, among high-risk HIV-negative transgender feminine, transgender masculine, and gender non-conforming youth and young adults for reducing sexual risk behaviors and increasing pre-exposure prophylaxis (PrEP) uptake. Participants are randomized into one of three conditions for a 6-month intervention: Group 1: culturally relevant theory-based text messages (Text+Step); or, Group 2: culturally relevant mobile-enhanced website (WebApp+Step); or, Group 3: informational website control condition with no theoretically based text messages or WebApp.

DETAILED DESCRIPTION:
TechStep is a three-arm, technology-based randomized controlled trial (RCT), with a stepped care approach, among high-risk HIV-negative transgender feminine, transgender masculine, and gender non-conforming youth and young adults for reducing sexual risk behaviors and increasing PrEP uptake. Transgender youth and young adults are enrolled for 9 months in the RCT. During the RCT, 250 participants will be enrolled and randomized to either: (1) text messaging (n=83), (2) WebApp (n=83), or (3) an informational website control (n=83) condition. Participants will include HIV-negative youth and young adults (ages 15-24) who are self-identified transgender feminine, transgender masculine or gender non-conforming. Participants will be recruited from venues in Boston, Houston, Los Angeles, New York, and Philadelphia. There will be four data collection time points: baseline, 3-, 6-, and 9-month. Visits will be conducted in-person at the venues, online, or some combination of in person or online. An ACASI will be completed using online survey tools. An HIV test, sexually transmitted infection (STI) panel, urine screen for recent illicit drug use, and blood microsampling or dried blood spot, for those who report PrEP uptake, to verify PrEP adherence will be collected in-person at the participants local venue, or via mailed self-collection kits. Process data of each participant activity at each step of the intervention, as well as the control intervention, will be collected. The study aims to measure the effects of the information-only (Info) arm compared to a text messaging intervention (Text+Step) to a WebApp intervention (WebApp+Step) for reducing sexual risk behaviors and increasing PrEP uptake.

ELIGIBILITY:
Inclusion Criteria:

* Report vaginal or anal sex (either insertive or receptive; excluding sex toys) with another person in the previous 12 months;
* Confirmed negative HIV test;
* Availability to meet with research staff in person or online at either the Baylor College of Medicine (BCM) Adolescent Medicine Trials Unit in Houston, Children's Hospital of Philadelphia, Children's Hospital Los Angeles, the PRIDE Health Research Consortium in New York City, or the Fenway Institute in Boston
* Have a mobile device with short messaging service (SMS; i.e. "texting") and Internet access capabilities; and
* Read and speak English (since the intervention is built in English)

Exclusion Criteria:

* Does not report vaginal or anal sex (either insertive or receptive; excluding sex toys) with another person in the previous 12 months;
* Reactive or indeterminate HIV test;
* Unable to meet with research staff in person or online at either the Baylor College of Medicine (BCM) Adolescent Medicine Trials Unit in Houston, Children's Hospital of Philadelphia, Children's Hospital Los Angeles, the PRIDE Health Research Consortium in New York City, or the Fenway Institute in Boston
* Does not have a mobile device with SMS and Internet access capabilities;
* Unable to read and speak English (since the intervention is built and delivered in English)
* Unwilling or unable to comply with protocol requirements;
* Unable to understand the Informed Consent/Assent Form.

Ages: 15 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Participants will include youth and young adults who are self-identified trans feminine, trans masculine or gender non-conforming OR whose birth sex and current gender differ
Enrollment: 254 (Actual)
Dates: Start 2019-10-18 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Hightow-Wideman, MD, MPH, Study Chair — University of North Carolina; Travis Sanchez, DVM, MPH, Study Chair — Emory University; Cathy J Reback, PhD, Principal Investigator — Friends Research Institute, Inc.; Keith J Horvath, PhD, Principal Investigator — San Diego State University
Locations (5):
- United States (5):
  - Children's Hospital Los Angeles, Los Angeles, California
  - The Fenway Institute, Boston, Massachusetts
  - PRIDE Health Research Consortium at Hunter CUNY, New York, New York
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
The investigators will assure the timely release and sharing of data two years after the publication of the main trial findings from the final dataset. Study variables will be available; however, the investigators will protect the rights and privacy of human subjects by redacting all identifiers from the data set. The de-identified data from this project will be available through individual requests directed to the Principal Investigator.

REFERENCES:
- [Derived] Reback CJ, Cain D, Rusow JA, Benkeser D, Schader L, Gwiazdowski BA, Skeen SJ, Hannah M, Belzer M, Castillo M, Mayer KH, Paul ME, Hill-Rorie J, Johnson ND, McAvoy-Banerjea J, Sanchez T, Hightow-Weidman LB, Sullivan PS, Horvath KJ. Technology-Based Interventions, with a Stepped Care Approach, for Reducing Sexual Risk Behaviors and Increasing PrEP Initiation Among Transgender and Gender Expansive Youth and Young Adults. AIDS Behav. 2024 Dec;28(12):3956-3969. doi: 10.1007/s10461-024-04513-w. Epub 2024 Sep 20. PMID 39304589
- [Derived] Reback CJ, Rusow JA, Cain D, Benkeser D, Arayasirikul S, Hightow-Weidman L, Horvath KJ. Technology-Based Stepped Care to Stem Transgender Adolescent Risk Transmission: Protocol for a Randomized Controlled Trial (TechStep). JMIR Res Protoc. 2020 Aug 13;9(8):e18326. doi: 10.2196/18326. PMID 32788149

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A confirmed negative HIV test was required to enroll in the study. Participants who used a remote enrollment option were offered at-home STI testing which included an HIV test. Participants who did not return at least the HIV test portion of the kit were subsequently and retroactively ineligible for the study, withdrawn, and not considered randomized.
Period: Overall Study
Arm/Group | Information | Text+Step | WebApp+Step
Started | 85 | 82 | 87
3-month Follow-up | 73 | 78 | 77
6-month Follow-up | 67 | 71 | 67
Completed | 69 | 72 | 70
Not Completed | 16 | 10 | 17
Not completed — Withdrawal by Subject | 5 | 3 | 4
Not completed — Lost to Follow-up | 11 | 7 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Text+Step | WebApp+Step | Information | Total
Number analyzed (Participants) | 82 | 87 | 85 | 254
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.88 (2.08) | 21.21 (1.87) | 21.57 (1.83) | 21.22 (1.94)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  nonbinary (assigned female at birth) | 39 | 40 | 34 | 113
  nonbinary (assigned male at birth) | 13 | 7 | 13 | 33
  trans feminine | 5 | 7 | 8 | 20
  trans masculine | 25 | 33 | 30 | 88
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21 | 20 | 20 | 61
  Not Hispanic or Latino | 60 | 66 | 63 | 189
  Unknown or Not Reported | 1 | 1 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 3 | 5
  Asian | 7 | 7 | 11 | 25
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 7 | 7 | 4 | 18
  White | 46 | 51 | 47 | 144
  More than one race | 16 | 15 | 14 | 45
  Unknown or Not Reported | 5 | 6 | 6 | 17
Region of Enrollment [Number; unit: participants]
  United States | 82 | 87 | 85 | 254

OUTCOME MEASURES:

1. Primary Outcome: Condomless Intercourse Events
Description: Participants will report the frequency of condomless sexual intercourse events they have engaged in for the past 3 months at baseline and at each follow-up. The value of interest is the cumulative number of events over follow-up.
Time Frame: 9 Months
Measure: Mean (95% Confidence Interval); unit: Expected events
Arm/Group | Text+Step | WebApp+Step | Information
Number analyzed (Participants) | 82 | 87 | 85
Expected events | 3.14 [2.45 to 3.82] | 3.17 [2.59 to 3.74] | 3.68 [3.16 to 4.20]
Statistical Analysis 1: Comparison: Text+Step vs Information; Test type: Superiority; p = 0.141, Longitudinal Targeted Maximum Likelihood; Average treatment effect = -0.54, 95% CI 2-sided [-1.26 to 0.18]
Statistical Analysis 2: Comparison: WebApp+Step vs Information; Test type: Superiority; p = 0.123, Longitudinal Targeted Maximum Likelihood; Average treatment effect = -0.51, 95% CI 2-sided [-1.16 to 0.14]

2. Primary Outcome: Condomless Intercourse Events While High on Drugs/Alcohol
Description: Participants will report the number of condomless sexual intercourse events they have engaged in while high on drugs or alcohol during their three most recent sexual encounters in the past 3 months at baseline and at each follow-up. The value of interest is the cumulative number of events over follow-up.
Time Frame: 9 Months
Measure: Mean (95% Confidence Interval); unit: Expected events
Arm/Group | Information | Text+Step | WebApp+Step
Number analyzed (Participants) | 85 | 82 | 87
Expected events | 1.04 [0.74 to 1.33] | 0.79 [0.55 to 1.04] | 1.02 [0.74 to 1.29]
Statistical Analysis 1: Comparison: Information vs Text+Step; Test type: Superiority; p = .127, Longitudinal Targeted Maximum Likelihood; Average treatment effect = -0.24, 95% CI 2-sided [-.56 to .07]
Statistical Analysis 2: Comparison: Information vs WebApp+Step; Test type: Superiority; p = .899, Longitudinal Targeted Maximum Likelihood; Average treatment effect = -.02, 95% CI 2-sided [-.34 to .30]

3. Primary Outcome: Condomless Intercourse Events During Sex Work
Description: Participants will report the number of exchange partners in the past 3 months at baseline and at each follow-up. The value of interest is the cumulative number of events over follow-up.
Time Frame: 9 Months
Population: Participants who answered the relevant survey questions necessary to assess the 3-month step-up criteria were included in the analytical sample.
Measure: Mean (95% Confidence Interval); unit: Expected events
Arm/Group | Information | Text+Step | WebApp+Step
Number analyzed (Participants) | 75 | 78 | 77
Expected events | 0 [0 to 0] | 0.03 [0.00 to 0.10] | 0 [0 to 0]

4. Primary Outcome: HIV Seroconversion
Description: HIV tests will be collected at each time point. Incident infections will be recorded.
Time Frame: 9 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Information | Text+Step | WebApp+Step
Number analyzed (Participants) | 85 | 82 | 87
Participants | 0 | 0 | 0

5. Primary Outcome: Incident STIs
Description: Participants will be tested for gonorrhea and chlamydia via throat, rectal, and urogenital swab specimen collection, as well as via urine samples at each time point. Incident STIs will be recorded.
Time Frame: 9 Months
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: Expected infections
Arm/Group | Information | Text+Step | WebApp+Step
Number analyzed (Participants) | 75 | 78 | 77
Expected infections | 0.06 [0 to 0.16] | 0.02 [0 to 0.07] | 0.04 [0 to 0.14]

ADVERSE EVENTS:
Time Frame: 9 months
Arm/Group | Information | Text+Step | WebApp+Step
All-Cause Mortality (participants affected / at risk) | 0/85 | 0/82 | 0/87
Serious Adverse Events (participants affected / at risk) | 0/85 | 0/82 | 0/87
Other Adverse Events (participants affected / at risk) | 2/85 | 1/82 | 3/87
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Information (N=85) | Text+Step (N=82) | WebApp+Step (N=87)
Unrelated mental health issues (Psychiatric disorders) | 2 | 0 | 1
Protocol related mental health concern (Psychiatric disorders) | 0 | 0 | 2
COVID (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-07-16): https://cdn.clinicaltrials.gov/large-docs/24/NCT04000724/Prot_SAP_000.pdf
  • Informed Consent Form (2021-02-24): https://cdn.clinicaltrials.gov/large-docs/24/NCT04000724/ICF_001.pdf